CLINICAL TRIAL: NCT03593187
Title: A Phase I/II Study of the Safety of CD34+ Haematopoietic Stem/Progenitor Cells and CD4+ T Lymphocytes Transduced With LVsh5/C46, a Dual Anti-HIV Gene Transfer Construct, in HIV-1 Infected Patients With High-risk Lymphoma
Brief Title: A Study Evaluating the Safety of Cal-1 (LVsh5/C46) Drug Product in HIV-1 Infected Patient With High Risk Lymphoma
Acronym: GENHIV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: CSL Behring (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P 141004; 2015-004453-41 (EudraCT Number)
Record Dates: First submitted 2018-06-15; First posted 2018-07-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: HIV-1 Infection
Keywords: HIV-1; Lymphoma; Gene therapy
MeSH Terms: conditions — Lymphoma | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cal-1( LVsh5/C46) drug product (Experimental)
  Interventions: Drug: Cal-1 (LVsh5/C46) drug product

INTERVENTIONS:
Drug: Cal-1 (LVsh5/C46) drug product — Autologous CD34+ Haematopoietic Stem/Progenitor Cells and CD4+ T Lymphocytes Transduced with LVsh5/C46, a Dual Anti-HIV Gene Transfer Construct

SUMMARY:
The purpose of this study is to evaluate the safety and the feasibility, and the success of engraftment of the introduction of Cal-1 gene-transduced haematopoietic cell populations (Ttn and HSPCtn) in patients with HIV-1-related high-risk lymphoma.

DETAILED DESCRIPTION:
not provided

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects will undergo screening assessments at three time points:

* Screening 1 at the beginning of chemotherapy,
* Screening 2 (first "check-point") after the harvest for CD34,
* Screening 3 (second "check-point") before the ASCT procedure. Potential subjects must satisfy all of the inclusion criteria to be enrolled in the study and proceed with the first apheresis (day -39).

In-A. Prior to any study-related procedures, signed informed consent indicating that they understand the purpose, risks and procedures required for the study and are willing to participate in the study In-B. Individuals aged 18 to 60 years of age (inclusive) at time of consent In-C. Women with child-bearing potential must be on adequate effective contraception (continuous progestative contraception) In-D. Documented HIV-1 infection at or before the time of lymphoma diagnosis In-E. Treatment with antiretroviral agents (excluding NNRTI) introduced or optimized at the time of screening

In-F. Biopsy-proven lymphoma meeting one of the following criteria:

1. 1. Intermediate- or high-grade B-cell non-Hodgkin lymphoma, meeting 1 of the following criteria:

   * in first complete remission with high-risk features such as T-cell lymphoma and plasmablastic lymphoma (after multidisciplinary consultation regarding the indication of ASCT in this context). The decision of ASCT is independent of the present clinical trial.
   * in partial remission
   * relapsed after initial complete remission
   * failed induction therapy but responds to salvage therapy (i.e., chemosensitive disease)
2. Hodgkin lymphoma, meeting 1 of the following criteria:

   * in first or greater relapse after initial complete remission
   * in partial remission
   * failed induction therapy but responds to salvage therapy (i.e. chemosensitive disease)
3. High-risk lymphoma requiring a treatment with combined chemotherapy and autologous stem cell transplantation (ASCT)

Exclusion Criteria:

Ex-A. -Left ventricular ejection fraction <50% at Screening 1:

Ex-B. Abnormal biochemistry at Screening 1:

Alanine and/or aspartate aminotransferase (ALT/AST) >10 x upper limit of normal (ULN) Total bilirubin > 2.5 x ULN Creatinine clearance <60ml/min Ex-C. Severe coagulopathy Ex-D. Prothombin time > 2x ULN Ex-E. Evidence of co-infection with hepatitis B virus (HBsAg+), hepatitis C virus, West Nile Virus, or Human T-lymphotropic virus (HTLV-1) as detected at Screening 1 Ex-F. Stay in West Nile Virus endemic area less than 6 weeks prior to CD34+ collection Ex-G. Evidence of non-treated opportunistic infection during the pre-infusion period Ex-H. Evidence of not-treated CNS involvement of lymphoma at Screening 1 Ex-I. Isolated CNS relapse of the lymphoma without other evidence of active disease at Screening 1 Ex-J. Known hypersensitivity to G-CSF (Neupogen™) or plerixafor (Mozobil™) Ex-K. Evidence of uncontrolled HIV-1 viremia at screening 2 and/or 3 (plasma HIV-1 RNA ≥ 1.000 copies/ml confirmed in 2 successive blood samples) Ex-L. Evidence of chemoresistant lymphoma at screening 2 Ex-M. Any contra-indication to ASCT at any time during the pre-infusion period Ex-N. Participation in any study involving any investigational drug or medical device within 3 months prior to Screening 1 Ex-O. Receipt of a vaccine for HIV-1 or any gene transfer product at any time Ex-P. Subjects who will not accept transfusions of blood products Ex-Q. Pregnant or breast-feeding woman at any time Ex-R. Woman of child-bearing potential not under adequate contraceptive protection at any time Ex-S. Inability to understand and provide informed consent Psychological or psychiatric disability thought to be clinically significant in the opinion of the investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse event post transplant | 24 months post-transplant
  to evaluate the procedure safety
Success of hematopoietic stem cell engraftment | 24 months post-transplant
  evaluation of Cal-1 marking and expression in peripheral blood subpopulations (monocytes, CD4+ and CD8+ lymphocytes)

SECONDARY OUTCOMES:
Overall survival | 24 months post-transplant
Absence of detection of vector-derived Replication competent lentivirus (RCL) | 24 months post-transplant
Frequency and severity of clinical adverse events | 24 months post-transplant
  as assessed by the United States national Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Absence of tropism shift from R5 to dual/mixed or X4 at any point after Day 0 | 24 months post-transplant
Quantify gene transfer efficiency and expression | 24 months post-transplant
  extent of HSPCtn and Ttn survival as measured by Cal-1 marking and expression in peripheral blood
Time to restart antiretroviral therapy | 24 months post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Marina CAVAZZANA, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Eric OKSENHENDLER, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Saint Louis, Paris, France

IPD SHARING:
Plan to Share IPD: No